CLINICAL TRIAL: NCT05609240
Title: Colo-Pro_2: A Feasibility Randomised Controlled Double Blind Trial to Compare Standard Bolus Dosed Cefuroxime Prophylaxis to Bolus-continuous Infusion Dosed Cefuroxime Prophylaxis for the Prevention of Infections After Colorectal Surgery
Brief Title: Colo-Pro_2: Bolus-continuous Infusion Cefuroxime Prophylaxis for the Prevention of Infections After Colorectal Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Birmingham (Other); Aneurin Bevan University Health Board (Other)
Responsible Party: Principal Investigator, Andrew Kirby, Associate Clinical Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 315251
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Antibiotic Prophylaxis; Colorectal Surgery
Keywords: Cefuroxime; Antibiotic; Colorectal; Prophylaxis; Surgery
MeSH Terms: interventions — Cefuroxime; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An anaesthetist will provide the intra-operative intervention and will the subsequently not be involved in the patients follow up or outcome assessment. alternatively, a research nurse not involved in participant follow up will provide the intra-operative intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Active Comparator): Cefuroxime 1.5 grams intravenous Administered in the hour before surgery and then 4 hourly intra-operatively.
  Interventions: Drug: Cefuroxime
- Intervention treatment (Active Comparator): Cefuroxime loading dose of 2332mg intravenous Administered in the hour before surgery.
  Following the loading dose a renal function based dosing will be given as a continuous intravenous infusion throughout surgery, as below. Continuous infusion will continue for up to 6 hours when it will return to 4 hourly dosing of cefuroxime at 1.5 grams intravenously, if required.
  Creatinine clearance (ml/min) and Cefuroxime:Dose per hour (mg/hr) 40-50ml/min=723mg/hr 50-60ml/min=867mg/hr 60-70ml/min=1011mg/hr 70-80ml/min=1155mg/hr >80ml/min=1227mg/hr
  Interventions: Drug: Cefuroxime

INTERVENTIONS:
Drug: Cefuroxime — See arm/group description
  Other Names: Cefuroxime sodium for injection

SUMMARY:
After a surgical operation patients may have an infection in the operation wound, the bladder, kidneys or lungs. To stop these infections patients are given a dose of antibiotic before their operation. Unfortunately, the amount of antibiotic available to fight infections falls throughout an operation, being removed from the body by the kidneys. Therefore, antibiotic levels may not be high enough to stop infections. A way of maintaining antibiotic levels throughout an operation is to give a single dose of antibiotic and then a constant amount of antibiotic by an infusion from the start to the end of the operation. A small single centre test study was previosuly undertaken into antibiotic dosing during bowel operations. One group of patients had a single dose of antibiotic before their operation. The other group had a single dose plus a constant dose of antibiotic until the end of their operation. The project showed patients were happy to take part and that the study was safe. The study helped us identify the correct amounts of antibiotic needed for the patients given the single dose plus a constant dose of antibiotic. This study was conducted at one hospital only, and wasn't big enough to confirm if one treatment was better than another or if results would be similar in other hospitals.

This study will build on the pilot study in a larger feasibility trial, the Colo-Pro_2 trial. It will be run in three hospitals so can assess if the trial design works at different hospitals. We will see if the results suggest one treatment, single dose of antibiotics before an operation, or single dose plus a constant dose of antibiotics throughout an operation, is better. This study will include up to 180 patients having bowel operations as they have a high risk of infection. All patients will be given the same antibiotic which is called cefuroxime. Cefuroxime is already used to stop infections after surgery. Using the same antibiotic in all patients means it is possible to know if differences in the number of infections are due to how the antibiotic is given. The number of infections that happen up to 30 days after operations will be counted. Staff looking after patients after the operation and those counting the infections will not know, unless necessary, the treatment patients received. This means the results won't be influenced by knowledge of the treatment received.

DETAILED DESCRIPTION:
See attached protocol

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective colorectal surgery (incision, excision or anastomosis of the large bowel, including anastomosis of small to large bowel)
* Age >16.
* Expected duration of surgery > 2hours
* Creatinine clearance > 40 ml/min
* Cefuroxime/metronidazole are appropriate antibiotic prophylaxis regimens.
* Patient capable of giving informed consent
* Patients undergoing colorectal surgery plus additional surgery e.g. plastic surgery, urological surgery, gynaecological surgery.

Exclusion Criteria:

* Unable to consent
* Pregnancy
* Expected duration of surgery <2hours
* Creatinine clearance <40ml/min
* Individual level microbiological advice for non-cefuroxime based prophylaxis
* Cephalosporin allergy
* Penicillin allergy (hypersensitivity reaction only)
* Coumarin (warfarin and acenocoumarol) treatment
* Seizure history or epilepsy
* Concurrent use of probenecid
* Current participation in a research project aimed at reducing surgical site infections (SSIs)
* Antibiotics for treatment of a systemic Gram negative infection within 12 hours of initiation of surgery (Vancomycin, Teicoplanin, Daptomycin, Linezolid, Flucloxacillin. Nitrofurantoin and Clarithromycin would be permissible antibiotics without systemic Gram negative antibiotics).
* A current diagnosis of infection at the time of study entry.
* STARR procedures (stapled trans anal resection of the rectum)
* Weight <30kg or >110kg

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 24 months
  Rate of recruitment
Retention rates | 90 days
  Rate of retention

SECONDARY OUTCOMES:
Health Care Associated Infection | 30 days
  The number of patients within 30 days of surgery with post-operative Health Care Associated Infection (HCAI). This will be defined by post-operative (> 72 hours) evidence of inflammation (fever, neutrophilia, C-Reactive Protein >100mg/L and infection (≥5 days prescription of antibiotic therapy) or bacteraemia with a recognised pathogen i.e., not a contaminant namely coagulase negative staphylococcus, Corynebacterium or Propionibacterium.
Surgical site infection | 30 days
  Superficial, deep and organ space surgical site infection. A wound assessment will be made at day 5 after operation and a questionnaire will be completed at day 30.
Microbiological evidence of urinary tract infection (UTI) | 30 days
  A urine sample with the detection of E.coli (or other Enterobacterales including Klebsiella, Enterobacter, Serratia, Citrobacter and Proteus)
Antimicrobial consumption after colorectal surgery | 90 days
  A day on which any antibiotic was consumed by a participant within 90 days of operations. Antibiotic prophylaxis e.g., for urinary tract infection, or splenectomy, are not included.
Antimicrobially resistant infections (AMR infections): | 90 days
  Infection with an antibiotic resistant bacteria will be identified by the rate of bacteraemia with the following antibiotic resistant bacteria detected in the blood stream:
  * Methicillin resistant Staphylococcus aureus
  * Vancomycin resistant Enterococcus faecalis/faecium
  * Extended spectrum beta-lactamase (ESBL) E.coli (or other Enterobacterales including Klebsiella, Enterobacter, Serratia, Citrobacter and Proteus
  * Carbapenemase producing Enterobacteriaceae (CPE) E.coli (or other Enterobacterales including Klebsiella, Enterobacter, Serratia, Citrobacter and Proteus)
C. difficile infection | 90 days
  A diagnosis of C. difficile infection (CDI) is one that requires confirmation of C. difficile toxin on a faeces test. Detection of the toxin gene by molecular testing is not sufficient. If multiple episodes if CDI infection, please report only the first episode
Anastomotic leakage after colorectal surgery | 90 days
  Radiological or surgical evidence of anastomotic leak
Mortality | 90 days
  Death
Length of hospital stay | 90 days
  The number of nights spend as a hospital in-patient within 90 days of operation.
Re-admission | 90 days
  Readmission to hospital following discharge with at least one night spent as a hospital in-patient.
Cost of healthcare treatment | 90 days
  Cost of healthcare treatment including days in hospital, surgical procedures and radiological procedures

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kirby, Study Chair — The Univeristy of Leeds
Locations (3):
- United Kingdom (3):
  - TheUniversity of Birmingham, Birmingham, West Midlands
  - Leeds Teaching Hospitals, Leeds, West Yorkshire
  - Aneurin Bevan University Health Board, Newport

IPD SHARING:
Plan to Share IPD: No